CLINICAL TRIAL: NCT05186259
Title: Modulating Mechanisms in Patients With Chronic Subjective Tinnitus and/or Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Bijzonder onderzoeksfonds (BOF) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BC-07036
Record Dates: First submitted 2021-11-24; First posted 2022-01-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Tinnitus; Pain
MeSH Terms: conditions — Tinnitus; Pain | interventions — Audiometry; Pain Measurement; Listening Effort

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with chronic tinnitus (Active Comparator): Patients with chronic subjective tinnitus (> 3 months)
  Interventions: Diagnostic Test: Self-reported signs of central sensitization; Diagnostic Test: Objective signs of central sensitization; Diagnostic Test: Audiological outcome measures (audiometry, tinnitus analysis, uncomfortable loudness) in tinnitus patients with and without pain; Diagnostic Test: Cognitive functioning; Diagnostic Test: Listening effort; Diagnostic Test: Self-reported psychological factors; Diagnostic Test: Self-reported lifestyle factors; Diagnostic Test: Self-reported quality of life; Diagnostic Test: Self-reported tinnitus severity and impact on daily life; Diagnostic Test: Self-reported hyperacusis; Diagnostic Test: Self-reported tinnitus characteristics
- Patients with chronic idiopathic neck pain (Active Comparator): Patients with chronic idiopathic neck pain (> 3 months)
  Interventions: Diagnostic Test: Self-reported signs of central sensitization; Diagnostic Test: Objective signs of central sensitization; Diagnostic Test: Self-reported psychological factors; Diagnostic Test: Self-reported lifestyle factors; Diagnostic Test: Self-reported measure of pain processing; Diagnostic Test: Self-reported quality of life; Diagnostic Test: Self reported neck pain related disability
- Patients with chronic tinnitus and chronic musculoskeletal pain (Active Comparator): Patients with chronic tinnitus and chronic musculoskeletal pain (> 3 months)
  Interventions: Diagnostic Test: Self-reported signs of central sensitization; Diagnostic Test: Objective signs of central sensitization; Diagnostic Test: Audiological outcome measures (audiometry, tinnitus analysis, uncomfortable loudness) in tinnitus patients with and without pain; Diagnostic Test: Cognitive functioning; Diagnostic Test: Listening effort; Diagnostic Test: Self-reported psychological factors; Diagnostic Test: Self-reported lifestyle factors; Diagnostic Test: Self-reported measure of pain processing; Diagnostic Test: Self-reported quality of life; Diagnostic Test: Self-reported tinnitus severity and impact on daily life; Diagnostic Test: Self-reported hyperacusis; Diagnostic Test: Self-reported tinnitus characteristics; Diagnostic Test: Self reported neck pain related disability
- Healthy controls (Active Comparator): Healthy controls without tinnitus or pain complaints
  Interventions: Diagnostic Test: Self-reported signs of central sensitization; Diagnostic Test: Objective signs of central sensitization; Diagnostic Test: Self-reported psychological factors; Diagnostic Test: Self-reported lifestyle factors; Diagnostic Test: Self-reported quality of life

INTERVENTIONS:
Diagnostic Test: Self-reported signs of central sensitization — Self-reported signs of central sensitization by means of the Central Sensitization Inventory (questionnaire)
Diagnostic Test: Objective signs of central sensitization — Objective signs of central sensitization by means of Quantitative Sensory Testing (mechanical and heat detection and pain thresholds, endogenous pain facilitation and inhibition)
Diagnostic Test: Audiological outcome measures (audiometry, tinnitus analysis, uncomfortable loudness) in tinnitus patients with and without pain — * Audiometry Performance of pure tone audiometry according to the modified Hughson-Westlake method
  * Tinnitus analysis Measurement of psychoacoustic features of tinnitus, including (1) tinnitus pitch, (2) loudness, (3) masking ability, and (4) residual inhibition.
  * Uncomfortable Loudness measures Performance of Uncomfortable Loudness measurements to evaluate the presence of hyperacusis. .
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Cognitive functioning — Evaluation of cognitive functioning by means of:
  * Auditory Stroop test
  * Detecting letters task
  * Letter-number sequencing task
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Listening effort — Evaluation of listening effort by means of the modified version of the behavioral listening effort test based on a dual-task paradigm by Degeest, Keppler & Corthals (2018) .
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Self-reported psychological factors — Evaluation of psychological factors by means of:
  * Depression, Anxiety and Stress Scale (DASS-21)
  * Beck Depression Inventory (BDI)
  * Big Five Inventory (BFI)
  * Connor-Davidson Resilience Scale
Diagnostic Test: Self-reported lifestyle factors — Evaluation of lifestyle factors by means of:
  Baecke Questionnaire Pittsburg Sleep Quality Index Insomnia Severity Index Stress subscale of the DASS 21
Diagnostic Test: Self-reported measure of pain processing — Evaluation of self-reported pain processing by means of the Pain Catastrophizing Scale
  Arms: Patients with chronic idiopathic neck pain; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Self-reported quality of life — Self-reported quality of life by means of the SF-36 questionnaire
Diagnostic Test: Self-reported tinnitus severity and impact on daily life — Evaluation of self-reported tinnitus severity and impact on daily life by means of the Tinnitus Functional Index
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Self-reported hyperacusis — Evaluation of self-reported characteristics of hyperacusis by means of the Hyperacusis Questionnaire
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Self-reported tinnitus characteristics — Evaluation of self-reported tinnitus characteristics by means of the Tinnitus Sample Case History Questionnaire
  Arms: Patients with chronic tinnitus; Patients with chronic tinnitus and chronic musculoskeletal pain
Diagnostic Test: Self reported neck pain related disability — Evaluation of self-reported neck pain related disability using the Neck Disability Index
  Arms: Patients with chronic idiopathic neck pain; Patients with chronic tinnitus and chronic musculoskeletal pain

SUMMARY:
This is a cross-sectional investigation into modulating mechanisms in patients with chronic subjective tinnitus, which will compare 4 patient groups namely chronic tinnitus with chronic pain, chronic tinnitus without chronic pain, chronic pain without tinnitus and healthy controls.

DETAILED DESCRIPTION:
The first aim is to investigate differences in pain-related factors, psychological factors, lifestyle factors and tinnitus-related factors in patients with chronic subjective tinnitus and the comparison with patients suffering from both chronic subjective tinnitus and chronic musculoskeletal pain, chronic musculoskeletal pain only and healthy controls. The primary outcome measures will be pain-related factors and correlations will also be calculated between pain-related factors on the one hand and psychological factors, lifestyle factors and tinnitus-related factors on the other hand.

A second aim is to assess contributing factors to tinnitus severity (measured by the Tinnitus Functional Index) in patients with tinnitus with or without chronic pain. Contributing factors will include pain-related factors, psychological factors, lifestyle factors, and tinnitus-related factors, audiological factors, cognitive factors.

* Pain-related factors include:

  1. Self-perceived symptoms of central sensitization by means of the Central Sensitization Inventory: The Central Sensitization Inventory is a self-report questionnaire that assesses clinical symptoms indicative for central sensitization.
  2. Experimental measures of central sensitization: Quantitative Sensory Testing Quantitative Sensory Testing (QST) is a psychophysiological assessment of sensory pathways including mechanicaldetection and pain thresholds, cutaneous heat detection and pain thresholds, and endogenous pain facilitation and inhibition.
  3. Self-reported pain processing by means of the Pain Catastrophizing Scale
  4. Self-reported neck pain related disability by means of the Neck Disability Index
* Psychological factors include:

Self-reported stress, anxiety and depression (Depression, Anxiety and Stress Scale_21 and Beck Depression Inventory), resilience (Connor Davidson Resilience Scale), personality (Big Five Index)

*Lifestyle factors include:

Self-reported physical activity (Baecke Questionnaire), self-reported sleep quality (Pittsburgh Sleep Quality Index) and self-reported insomnia severity (Insomnia Severity Index), self-reported quality of life (SF-36)

*Tinnitus-related factors include:

Self-reported tinnitus severity and impact (Tinnitus Functional Index), self-reported hyperacusis (Hyperacusis Questionnare), self-reported tinnitus characteristics (Tinnitus Sample Case History Questionnaire)

* Cognitive factors include:

  1. Verbal working memory capacity and processing speed (Letter-number sequencing task)
  2. Attention span (detecting letters-task (COTESS))
  3. Cognitive flexibility and inhibition (Auditory Stroop task)
  4. Listening effort (Modified version of the behavioral listening effort test based on a dual-task paradigm by Degeest, Keppler & Corthals (2018))
* Audiological factors include:

  1. Hearing thresholds (Pure tone audiometry)
  2. Psychoacoustic features of tinnitus (tinnitus pitch, loudness, masking ability, and residual inhibition using same devices as for pure tone audiometry)
  3. Uncomfortable Loudness (using same devices as for pure tone audiometry)

ELIGIBILITY:
Inclusion Criteria:

* Chronic subjective tinnitus patients without chronic pain:

  * Aged between 18-65 years
  * Chronic subjective tinnitus (> 3 months during most of the days (4 or more)and for more than 5 minutes/day)
  * Speaking and understanding Dutch fluently
* Chronic subjective tinnitus patients with chronic pain:

  * Aged between 18-65 years
  * Chronic subjective tinnitus (> 3 months during most of the days (4 or more)and for more than 5 minutes/day)
  * Speaking and understanding Dutch fluently
  * Persistent musculoskeletal pain lasting more than 3 months
  * Mean pain intensity of more than 3 of 10 on a numeric pain rating scale during the preceding month (the cutoff for clinically relevant pain)
* Chronic ideopathic neck pain:

  * Aged between 18-65 years
  * Persistent neck pain lasting more than 3 months
  * Mean pain intensity of more than 3 of 10 on a numeric pain rating scale during the preceding month (the cutoff for clinically relevant pain)
* Healthy controls:

  * Aged between 18-65 years

Exclusion Criteria:

* Chronic subjective tinnitus with/without chronic pain:

  * Objective tinnitus
  * Subjective tinnitus caused by clear causes such as tumor, trauma, vascular dysfunction, neurological disorder, pulsatile tinnitus
  * Vertigo (Menière's disease, BPPV,…)
  * Deafness
  * Progressive middle ear pathology
  * Intracranial pathologies
  * Subjects with prior otologic surgery (for example stapedotomy), active outer or middle ear pathology
  * History of head, neck or shoulder trauma or surgery (< 5 years, or remaining complaints)
  * A history of whiplash trauma
  * Major depression or psychiatric illness (diagnosed by a psychiatrist and being in medicamental or psychiatric treatment)
  * Life threatening, metabolic, cardiovascular, neurologic, systemic diseases
  * Diagnosis of fibromyalgia/chronic fatigue syndrome
  * Pregnancy or given birth in the preceding year
  * Dyslexia, dyscalculia, AD(H)D, language/communication disorder
* Chronic subjective tinnitus without chronic pain (additional exclusion criteria):

  * No history of chronic pain
  * No pain condition in the last 6 months for which treatment was sought
  * No pain in any region > 2/10 on the testing day
* Chronic ideopathic neck pain:

  * Ever experienced whiplash trauma or other form of trauma to the head, neck, or upper quadrant
  * Specific causes of neck pain, such as cervical hernias with clinical symptoms
  * Major depression or psychiatric illness (diagnosed by a psychiatrist and being in medicamental or psychiatric treatment)
  * Life threatening, metabolic, cardiovascular, neurologic, systemic diseases
  * Diagnosis of fibromyalgia/chronic fatigue syndrome
  * A history of neck, head or shoulder girdle surgery
  * A history of whiplash trauma
  * Pregnancy or given birth in the preceding year
  * Diagnosis of any TMD, according to the Research Diagnostic Criteria for TMD (RDC/TMD); or concomitant diagnosis of primary headache
* Healthy controls:

  * Any form of tinnitus and/or hyperacusis
  * Experiencing any type of pain during at least 8 consecutive days with an NRS higher than 2/10 in the preceding year
  * Reported pain on the day of testing (VAS higher than 2/10)
  * Vertigo (Menière's disease, BPPV,…)
  * Deafness
  * History of head, neck or shoulder trauma or surgery (< 5 years, or remaining complaints)
  * Wearing a hearing aid device, implant, noise generators or receiving neuromodulation therapy
  * Intracranial pathologies
  * History of head, neck or shoulder trauma or surgery (< 5 years, currently no complaints)
  * Major depression or psychiatric illness (diagnosed by a psychiatrist and being in medicamental or psychiatric treatment)
  * Life threatening, metabolic, cardiovascular, neurologic, systemic diseases
  * A history of whiplash trauma
  * Diagnosis of fibromyalgia/chronic fatigue syndrome
  * Pregnancy or given birth in the preceding year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Between-group differences in mechanical pain sensitivity by means of pressure detection and pain thresholds (expressed in kgf) | At baseline
  Pain sensitivity will be assessed by a mechanical stimulus, which is given by the tester with a digital pressure algometer (FDX; Wagner Instruments) at a rate of 1 kg pressure rise per second. The participant is asked to say 'yes' if the point was reached when the pressure stimulus causes a sensation of pain (detection threshold), the tester continues giving pressure until the patient says 'yes' for a second time indicating the feeling of pain reached a 6/10 of the NRS (pain threshold). T Two consecutive measurements with a break of 30 seconds are performed.
  This protocol is performed at 5 standardized body locations, being: C5-C cervical joint, N. Trigeminus, M. Masseter, M. Extensor carpi radialis longus, M. Tibialis Anterior

SECONDARY OUTCOMES:
Tinnitus analysis | At baseline
  Tinnitus analysis Psychoacoustic features of tinnitus will be determined using the same equipment that was used for pure tone audiometry. The tinnitus analysis included determining.
Audiometric assessments | At baseline
  Audiometry Pure tone audiometry according to the modified Hughson-Westlake method will be performed. For air conduction, pure tone thresholds will be determined at octave frequencies from 0.25 to 8 kHz and at half-octave frequencies 3 and 6 kHz (DD45 audiometric headset, Calisto audiometer, Interacoustics).
  For each ear separately, hearing thresholds (using tonal luminal audiometry) and uncomfortable loudness (UCL) levels were determined on all octave frequencies between 250 and 8000 Hertz (Hz). Based on the audiometric thresholds and UCL levels, the Johnson Hyperacusis Quotient.
Between-group differences in heat pain sensitivity by means of heat detection and pain thresholds (expressed in °) | At baseline
  Heat stimuli are given using the CHEPS PATHWAY system (Medoc). This probe is placed on the skin at the 5 standardized locations. It provides a heat stimulus that rises at a rate of 1°C/second.
  Using a dual response button, the participant has to indicate when the heat sensation changes into a pain sensation by pressing a blue button (detection threshold). The temperature keeps rising after the blue button is pressed. If the patient scores the pain sensation resulting from the heat stimulus as a 6/10 on the NRS they have to press the red button. At that moment, the temperature of the thermode goes back to the baseline temperature of 32°C. When the baseline temperature is reached, a second heat stimulus is given after a 15 second break. 3 consecutive trials will be performed.
  This protocol is performed at 5 standardized body locations, being: C5-C cervical joint, N. Trigeminus, M. Masseter, M. Extensor carpi radialis longus, M. Tibialis Anterior
Between-group differences in endogenous pain facilitation by means of a temporal summation protocol (expressed in pain scores (numeric rating scales, NRS) | At baseline
  Temporal Summation is performed with the Contact Heat-Evoked Potential Stimulator (CHEPS) model. Temporal summation is evaluated at the M. tibialis anterior and the M. extensor carpi radialis longus.
  The temperature corresponding with the mean score of the 6/10 NRS score (heat pain threshold) from the corresponding body part is used as the painful stimulus. Ten stimuli from the same heat are given to the participant with a thermode. After stimulus 1, 5 and 10 a beep sound is heard. At these moments the participant has to score the pain that they experience from the previous stimulus on the NRS from 0 to 10. Between stimuli the temperature goes back to the baseline temperature of 32°C. The velocity of the heating is 70°C/second and the velocity of the cooling down is 40°/second. Each stimulus is 0.5 seconds long with a frequency of 0.5 Hz.
Between-group differences in endogenous pain inhibition by means of conditioned pain modulation protocol (expressed in kgf and °) | At baseline
  Conditioned pain modulation is tested by asking the participant to put their non- non-dominant or non-painful dominant hand (up to the wrist joint) in a water bath of 45,5°C for 1 minute. This is the conditioning stimulus. After this, a PPT measurement is performed to measure pressure detection and pain thresholds again, at the level of the M. extensor carpi radialis longus. Two consecutive measurements of the PPTs are being performed with a 30 seconds interval in between. Thereafter, the non-dominant or non-painful hand is placed in the hot water for another minute and after this minute, heat detection and pain thresholds are evaluated again at the M. extensor carpi radialis longus. Both pressure and heat are the testing stimulus.
  Also, the NRS score (0-10) for the water was asked to know if they perceived the water as a high enough pain stimulus.
Between-group differences in self-reported signs of central sensitization by means of the Dutch version of the Central Sensitization Inventory (questionnaire) | At baseline
  The Central Sensitization Inventory measures the somatic and emotional symptoms commonly associated with central sensitization. It consists of two parts, one measuring 25 symptoms, the other asks whether patients have been previously diagnosed with ten specific diagnoses. A cut off of 40 out of 100 is used to determine the presence of self-reported signs of central sensitization (the higher the score, the higher the severity).
Between-group differences in self-reported psychological factors | At baseline
  Three negative emotional dimensions: 'depression', 'anxiety' and 'stress were evaluated using the self-report Depression Anxiety and Stress Scale 21 (DASS21), which is a short version of the DASS.The total score ranges between 0 and 126 and higher scores indicate more severe negative emotional status.
Between-group differences in self-reported psychological factors | At baseline
  The Dutch version of the Beck Depression Inventory (BDI) was used for the assessment of depression. The total score of the BDI ranges between 0 and 63 and higher scores reflect more severe depression.
Between-group differences in self-reported psychological factors | At baseline
  The Dutch version of the Connor-Davidson Resilience Scale 25 (CD-RISC 25) was used to assess resilience, which is a measure of stress coping ability. The total score ranges between 0 and 100 and a higher score reflects greater resilience.
Between-group differences in self-reported psychological factors | At baseline
  The Big Five Index 2 (BFI-2) was used to quantify five traits of personality, namely agreeableness, conscientiousness, extraversion, neuroticism, and openness. The BFI-2 consists of 15 facets, describing different features of each trait
Between-group differences in self-reported lifestyle factors | At baseline
  Self-reported physical activity levels were evaluated using the Baecke Physical Activity Questionnaire. This questionnaire consists of 16 items assessing three different domains of physical activity: work, sports and leisure time. The total score varies between 3 and 15 with a higher score reflecting a greater level of physical activity.
Between-group differences in self-reported lifestyle factors | At baseline
  The Pittsburgh Sleep Quality Index (PSQI) was used to evaluate self-perceived overall sleep quality in 7 domains: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, sleep medication, and daytime dysfunction over the previous month. The maximal score ranges between 0 and 21, and a global score of 5 or higher indicates clinically significant sleep problems
Between-group differences in self-reported lifestyle factors | At baseline
  The Insomnia Severity Index (ISI) was used to assess the patient's perception of insomnia severity. The ISI consists of seven items assessing the severity of sleep onset and sleep maintenance difficulties (both nocturnal and early morning awakenings), satisfaction with current sleep pattern, interference with daily functioning, notice ability of impairment attributed to the sleep problem and degree of distress or concern caused by the sleep problem. The maximal score ranges between 0 and 28 and higher scores indicate more severe insomnia.
Between-group differences in self-reported quality of life | At baseline
  Self-reported health-related quality of life will be evaluated using the SF- 36. This self-report questionnaire consists of 36 items that can be clustered into eight subscales: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. The summation of all subscales provides the total score (0-800).
Between-group differences in self-reported neck pain related measures | At baseline
  The Dutch version of the Neck Disability Index (NDI) will be used to evaluate the level of self-reported pain-related disability. The NDI consists of 10 items and has a total score of 50. Higher NDI scores reflect higher levels of neck pain-related disability. A score between 0 and 4 reflects no disability, a score between 5 and 14 indicates mild disability, between 15 and 24 moderate disability, between 25 and 34 severe disability and > 35 is considered as complete disability. (
Between-group differences in self-reported neck pain related measures | At baseline
  Neck pain catastrophizing will be assessed using the Dutch Pain Catastrophizing Scale (PCS), which is a self-report questionnaire to evaluate the presence of catastrophic thoughts and feelings towards pain. The PCS consists of 13 items and has a maximal score of 52. Higher scores indicate higher levels of pain catastrophizing. The PCS includes three subscales; magnification (experiencing pain as a threat), rumination (repeated worrying), and helplessness (believing that nothing can resolve the pain).
Between-group differences in self-reported tinnitus related measures | At baseline
  The Dutch validated version of the Tinnitus Sample Case History Questionnaire (TSCHQ) will be used for the standardized collection of information regarding the tinnitus history, tinnitus characteristics, modulating factors and other symptoms such as neck pain or headache.
Between-group differences in self-reported tinnitus related measures | At baseline
  The Dutch validated version of the Tinnitus Functional Index (TFI) will be used to evaluate tinnitus impact. The TFI is a 25-item self-report questionnaire with a total score ranging between 0 and 100, which consists of eight different subscales (intrusiveness, cognition, sleep, sense of control, relaxation, emotional, auditory and quality of life subscales). The higher the score, the higher the tinnitus impact.
Between-group differences in self-reported tinnitus related measures | At baseline
  The Dutch version of the Hyperacusis Questionnaire (HQ) will be used for the quantification and characterization of hyperacusis. The HQ consists of 14 items with a total score ranging between 0 and 42, a score greater than 28 is considered to represent auditory hypersensitivity or hyperacusis.
Cognitive functioning | At baseline
  The Auditory Stroop test will be used to measure cognitive flexibility and inhibition.
Cognitive functioning | At baseline
  The detecting letters-task (COTESS) will be used to test the participant's attention span.
Cognitive functioning | At baseline
  The letter-number sequencing task is part of the Wechsler Adults Intelligence Scale (WAIS-IV-NL) and will be used to evaluate verbal working memory capacity and processing speed.
Cognitive functioning | At baseline
  A modified version of the behavioral listening effort test based on a dual-task paradigm by Degeest, Keppler & Corthals (2018) will be used. The test consists of a primary and secondary task that will be administered separately (baseline condition) and simultaneously ( dual-task condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Meulemeester K, Meeus M, De Pauw R, Cagnie B, Keppler H, Lenoir D. Suffering from chronic tinnitus, chronic neck pain, or both: Does it impact the presence of signs and symptoms of central sensitization? PLoS One. 2023 Aug 24;18(8):e0290116. doi: 10.1371/journal.pone.0290116. eCollection 2023. PMID 37616265